CLINICAL TRIAL: NCT06683963
Title: AI-Assisted TelerehabiLitAtion System (ATLAS) for Post-discharge Continuation of Rehabilitative Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Community Hospitals (Other)
Collaborators: Rebee Health (Unknown); Jurong Community Hospital (Unknown)
Responsible Party: Principal Investigator, Low Lian Leng, A/Prof, SingHealth Community Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20242246
Record Dates: First submitted 2024-10-29; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Rehabilitation; Deconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control - usual care (No Intervention): Business as usual in community hospital, no added device intervention
- Intervention - Rebee (Experimental): Addition of Rebee device during and after community hospital stay
  Interventions: Device: Rebee

INTERVENTIONS:
Device: Rebee — Tablet device with accompanying sensor device. Tablet device is preloaded with exercises, to be taught to patients during their hospital stay, and to be continued post-discharge
  Arms: Intervention - Rebee

SUMMARY:
The study team proposes ATLAS (AI-Assisted TelerehabiLitAtion System) a two-part solution. The first-Rebee AI-assisted telerehabilitation device-assists in inpatient rehabilitation, and allows patients to continue with their physical rehabilitation when discharged and waiting for Day Rehabilitation Centre (DRC). The second-a structured programme to train and familiarise patients and caregivers to Rebee over patients' Community Hospital (CH) inpatient rehabilitation stay-adopts an evidence-based approach to increase uptake and adherence to Rebee.

ELIGIBILITY:
Inclusion Criteria:

1. Rehabilitation Diagnostic Group (RDG): Total Knee Replacement / Deconditioning
2. Age 60 and above
3. Speak English/Mandarin
4. Able to follow instructions, no cognitive impairment
5. No MDRO (MultiDrug Resistant Organism)
6. Suitable and able to wear motion sensor on upper and lower limbs
7. Suitable and able to engage in Rebee exercises

Exclusion Criteria:

1. Not under RDG: Total Knee Replacement / Deconditioning
2. Below 60 years old
3. Unable to speak English/Mandarin
4. Cognitive impaired, unable to follow instructions
5. Has MDRO
6. Not suitable to wear motion sensor on upper and lower limbs
7. Refusal to participate / give informed consent

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Barthel Index scores from baseline to 4, 8, and 12 weeks | from recruitment (week 0) till end of study at 12 weeks
  Modified Barthel Index (MBI) measures ability to complete activities of daily living (ADLs).
  Scores range from 0 to 100. A higher score represents more independence, a lower score indicates more assistance needed (ie less independent).
  0-20: Total dependence, 21-60: Severe dependence, 61-90: Moderate dependence, 91-99: Slight dependence, 100: Independence.

SECONDARY OUTCOMES:
Change in Quality of Life scores from baseline to 4, 8, and 12 weeks | from recruitment (week 0) till end of study at 12 weeks
  Quality of Life as measured using EQ-5D-5L.
  Has two components to this instrument:
  1. EQ-5D descriptive system
     * 1 to 5 for each dimension
     * A higher score represents "worse health status" (i.e., more severe problems with dimension).
  2. EQ visual analogue scale (EQ VAS)
     * 0 to 100
     * A higher score represents "better health status" (i.e., overall current health status).
Change in Patient Activation Level from baseline to 4, 8, and 12 weeks | from recruitment (week 0) till end of study at 12 weeks
  Patient Activation Level measured using PAM-13 Score from 0 to 100 Higher scores indicate greater patient activation
Readmission rates to hospital within 30 days of discharge | within 30 days from discharge date
  e.g. 0 means no readmissions back to hospital within 30 days of discharge occured
Change in Joint range of motion from baseline to 4, 8, and 12 weeks | from recruitment (week 0) till end of study at 12 weeks
  Measured Joint Range of operated knee for patients with total knee replacement (TKR) Joint range will be measured for knee Extension and well as knee Flexion
Length of Stay in Community Hospital reported in days | From recruitment (week 0) till end of study at 12 weeks
  Length of (inpatient) Stay in Community Hospital Reported in days, as measured by Discharge Date minus Admission Date e.g. if Discharge Date is 3/11/2024, and Admission Date is 1/11/2024, patient stayed for 2 days as an inpatient in the community hospital
Change in STS (sit to stand) score from baseline to 4, 8, and 12 weeks | from recruitment (week 0) till end of study at 12 weeks
  Time taken to Sit to Stand 5 times, calculated in seconds A higher score represents taking a longer time to complete 5 times sit to stand.

IPD SHARING:
Plan to Share IPD: No